CLINICAL TRIAL: NCT05728684
Title: A Single-arm Study Sponsored by Investigators to Evaluate the Efficacy and Safety of CM310 Recombinant Humanized Monoclonal Antibody Injection in Patients With Recurrent IgG4-related Diseases
Brief Title: Study to Evaluate the Efficacy and Safety of CM310 in Subjects With IgG4-related Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Liu Yanying, Deputy Director of Rheumatology Department, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YYXSSC-IIT-002
Record Dates: First submitted 2023-01-17; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: IgG4 Related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM310 (Experimental): CM310, subcutaneous
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — CM310 Injection

SUMMARY:
This study is a single-arm study initiated to evaluate the efficacy and safety of CM310 in subjects with recurrent IgG4-related disease.

DETAILED DESCRIPTION:
This study includes three stages: screening period, treatment period and safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years, male and female.
* With IGG4-related disease.

Exclusion Criteria:

* Inoculate live vaccine within 4 weeks before screening.
* Treponema pallidum antibody positive in screening period.
* Active hepatitis in screening period.
* With a history of solid organ or cell transplantation within 6 months before screening.
* With other medical or non-medical conditions that are not suitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Response rate | up to week 12
  Response rate after administration for 12 weeks